CLINICAL TRIAL: NCT03940638
Title: Management of Septic Non-union of the Tibia Using the "Induced Membrane" Technique
Acronym: SEPT-LEG
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao002
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Septic Tibial Non-union
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic non-union of the tibia
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
The aim of the study was to assess clinical and radiological results with the "induces membrane" technique, described by A. C. Masquelet in 1986, in a series of patients with septic non-union of the tibia

DETAILED DESCRIPTION:
Septic tibial non-union is a therapeutic challenge that may even lead to amputation. Treatment often necessitates several chirurgical steps. It is agreed that resection must extend to several tissues (osteitis zone ans macroscopically pathological soft tissue), with associated non-union site stabilization ans effective antibiotic therapy.

In 1986, Pr A. C. Masquelet described a 2-step procedure called the induced membrane technique, to manage bone defects of varying severity. Initial results were encouraging but there have been few large homogeneous series specific to this technique in septic non-union.

ELIGIBILITY:
inclusion criteria :

* Patients with septic non-union of the tibia
* managed using the induced membrane technique between novembrer 2007 and novembre 2014 in Reims University hospital
* Patients who agree to participate to the study
* Major patient

exclusion criteria :

* Patient under law protection
* Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic non-union of the tibia managed using the induced membrane technique
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Presence of Bone union | Day 0
  Bone union was defined by 2 continuous cortices on 2 views (radiologic images comprising 2 perpendicular views of the affected segment)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Siboni R, Joseph E, Blasco L, Barbe C, Bajolet O, Diallo S, Ohl X. Management of septic non-union of the tibia by the induced membrane technique. What factors could improve results? Orthop Traumatol Surg Res. 2018 Oct;104(6):911-915. doi: 10.1016/j.otsr.2018.04.013. Epub 2018 Jun 7. PMID 29886150